CLINICAL TRIAL: NCT01731288
Title: Pregnancy, Childbirth Intentions and Outcomes Under Sexual Pain
Acronym: PRECIOUS
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Other Study IDs: H11-00968
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Vulvodynia; Provoked Vestibulodynia
Keywords: pregnancy; childbirth; pain; vulvodynia; provoked vestibulodynia
MeSH Terms: conditions — Vulvodynia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- vulvodynia: Women with vulvodynia
- control: Women without vulvar pain

SUMMARY:
The main purpose of this study is to assess conception, pregnancy, childbirth, and pain experiences among women who have been diagnosed with vulvodynia. Specifically, this study aims to examine the following among women who have been diagnosed with vulvodynia: 1) rates of pregnancy/childbirth and desire for children; 2) fear of pregnancy and childbirth; 3) potential difficulties experienced while attempting to become pregnant and during pregnancy/childbirth; 4) methods used to become pregnant and deliver; 5) methods used to manage vulvodynia symptoms during pregnancy; and 6) pain outcomes associated with pregnancy.

Very little research has examined pregnancy/childbirth experiences among women with vulvodynia, or the natural history of vulvodynia. As such this is a preliminary investigation that will provide descriptive information regarding many of the proposed research questions. Based on the clinical experience of the investigators, it is expected that women with vulvodynia will report lower rates of pregnancy and higher levels of fear about pregnancy and childbirth in comparison to women without such pain. It is also expected that women with vulvodynia will report more difficulties becoming pregnant as compared to women without such pain, and that women with vulvodynia will report more elective nonvaginal births in comparison to vaginal births.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of vulvodynia from a physician (women with vulvodynia only)
* assessed and/or treated at one of 3 clinics (women with vulvodynia only)
* free from chronic vulvar pain and pain with sexual intercourse in their lifetime (control women only)
* 19 years of age or older
* fluent in English

Exclusion Criteria:

* younger than 19 years of age
* lack of fluency in English

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group consists of a community sample. The vulvodynia group consists of women who have been diagnosed with vulvodynia/provoked vestibulodynia and who have been assessed and/or treated at 1 of 3 tertiary clinics:
  1) Vulvar Pain Clinic (no longer active) located at the Women's Clinic, Willow Pavilion, Vancouver General Hospital; 2) Multidisciplinary Vulvodynia Program (MVP); or 3) BC Centre for Sexual Medicine
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rates | data is collected at a single time point
  We will assess if women with vulvodynia experience different rates of pregnancy in comparison to women without such pain
Intentions to have children | data is collected at a single time point
  We will assess how many women with vulvodynia wish to have children in their lifetime.
Fear of pregnancy/childbirth | data is collected at a single time point
  We will assess if women with vulvodynia report higher levels of fear about pregnancy and childbirth in comparison to women without such pain.
Difficulties becoming pregnant | data is collected at a single time point
  We will assess if women with vulvodynia experience more difficulties becoming pregnant in comparison to women without such pain.
Pregnancy/delivery complications | data is collected at a single time point.
  We will assess if women with vulvodynia experience more complications during pregnancy and delivery in comparison to women without such pain.
Pregnancy/delivery methods | data is collected at a single time point
  We will assess what methods women with vulvodynia use to become pregnant and deliver.
Symptom management during pregnancy | data is collected at a single time point
  We will assess how women manage their vulvodynia symptoms during pregnancy.
Change of pain symptoms during and after pregnancy | data is collected at a single time point
  We will assess if vulvodynia-related pain symptoms change during and after pregnancy.

SECONDARY OUTCOMES:
Course of vulvodynia | data is collected at a single time point
  We will assess the course of vulvodynia after treatment is received from health care workers specializing in vulvar pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Diamond Health Care Centre, Vancouver Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- See also: University of British Columbia Sexual Health Lab website — http://www.obgyn.ubc.ca/SexualHealth/